CLINICAL TRIAL: NCT06437392
Title: Evaluation of Sarcopenia and Related Factors in Patients Diagnosed With Psoriatic Arthritis
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gonca Canan Doğan Tosun, Medical Doctor (Physical Medicine and Rehabilitation), Ankara City Hospital Bilkent
Other Study IDs: 10026356
Record Dates: First submitted 2024-05-19; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Psoriatic Arthritis
Keywords: rheumatic disease; sarcopenia; ultrasonography
MeSH Terms: conditions — Arthritis, Psoriatic; Rheumatic Diseases; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriatic arthritis: Psoriatic arthritis patient
- Healthy volunteer: Healthy Volunteer

SUMMARY:
The purpose of the study is identify the prevalence of sarcopenia and its associated factors in patients with psoriatic arthritis. Furthermore, we aimed to investigate the predictive contribution of USG in diagnosing sarcopenia by assessing the thickness of the rectus femoris, vastus intermedius, and quadriceps muscles in patients with psoriatic arthritis.

DETAILED DESCRIPTION:
After being informed about study and potential risk, all patient and giving written informed consent will undergo screnneing determite eligibility for study entire. Participants who agree to take part in the study and sign the informed consent form will be divided into two groups: patients and healthy volunteers. The patients will undergo a rheumatological examination, and sarcopenia screening will be conducted for both groups. Additionally, the quadriceps muscle thickness of both groups will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with psoriatic arthritis according to CASPAR criteria at least 1 year ago
* Between 18 and 65 years old
* Normal cognitive functions
* Agrees to participate in the study
* No changes in medical treatment for psoriatic arthritis in the last 3 months

Exclusion Criteria:

* Those with neurological diseases
* Those with hip dysplasia
* Those with upper and lower extremity deformities
* Those with upper and lower extremity joint arthroplasty
* Those with arthritis and deformities in the hands
* Those with lumbar stabilization
* Those with cognitive impairment preventing participation in the study
* Those with body weight beyond the device's measurement capacity
* Those who do not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65, who were diagnosed with psoriatic arthritis at least one year ago according to the CASPAR criteria, and healthy controls, who visited Ankara Bilkent City Hospital Physical Medicine and Rehabilitation Department, were included.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 1 day
  muscle strength measurement:Hand grip strength is a parameter used to assess sarcopenia. Therefore, the hand grip strength of participants will be measured. A Jamar hydraulic hand dynamometer (FEI®, model 5030J1, USA) will be used for measuring muscle strength.For the hand grip strength measurement, participants will be seated with back support, with the shoulder in adduction, the elbow at 90 degrees flexion, the forearm and wrist in neutral and supported
4 m gait speed test | 1 day
  Participants are instructed to walk at a normal pace on a flat 6-meter surface (including the first 1 meter for acceleration, 4 meters for the walking test area, and the last 1 meter for deceleration). Those who take longer than 5 seconds to complete the 4 meters (walking speed <0.8 m/s) are evaluated as having low physical performance.
Quality of life in sarcopenia scale (SARQoL) | 1 day
  The SARQoL (Sarcopenia Quality of Life) questionnaire consists of 55 items and 22 questions, organized into seven different domains of quality of life: physical and mental health, locomotion, body composition, functionality, daily living activities, leisure activities, and fears.
Tinetti balance and walking test | 1 day
  It is a test that assesses the participants' balance and walking. It includes 9 questions for balance and 7 questions for walking. Each response is scored between 0 and 2 points.
Hospital Anxiety and Depression Scale | 1 day
  It is a scale developed to identify cases of anxiety disorders and depression in patients in non-psychiatric hospital clinics. Both contain seven intertwined items.
PSAID12 | 1 day
  This is a questionnaire that assesses the quality of life of patients diagnosed with psoriatic arthritis. It addresses pain, fatigue, skin problems, ability to perform work and/or leisure activities, functional capacity, discomfort, sleep disturbances, embarrassment from appearance, social participation, and depression.In this test, patients receive a score between 0 and 10.
DAS 28 | 1 day
  In the method where tenderness and swelling in 28 joints are recorded, known as the Disease Activity Score (DAS 28), global pain assessment score is used along with CRP (C-Reactive Protein) or ESR (Erythrocyte Sedimentation Rate) values. Scores of 2.6 or lower are considered remission, while scores between 2.6 and 3.2 indicate low disease activity, scores between 3.2 and 5.1 indicate moderate disease activity, and scores above 5.1 indicate high disease activity.
BASDAI | 1 day
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score consists of six questions in the form of a visual analog scale (VAS) related to the five main symptoms of Ankylosing Spondylitis over the past week: fatigue, spinal pain, peripheral joint pain/swelling, localized tenderness, and morning stiffness. A final score between 0 and 10 is obtained. A BASDAI score of 4 or higher is considered indicative of active disease.
DAPSA | 1 day
  The Disease Activity Index for Psoriatic Arthritis (DAPSA) score involves a joint examination of the patient. 68 joints are assessed for tenderness, and 66 joints for swelling. The numbers of tender and swollen joints are determined. The physician evaluates the patient's overall pain during examination and scores it out of 10. The patient's Visual Analog Scale (VAS) value is also recorded. The CRP value is noted.
  The score is then calculated simply by summing up all these values (number of tender joints + number of swollen joints + physician's assessment of overall pain + VAS + CRP).
  A score between 0 and 4 indicates remission, 5 to 14 indicates low disease activity, 15 to 27 indicates moderate disease activity, and a score greater than 28 indicates high disease activity.
PASI | 1 day
  The Psoriasis Area Severity Index (PASI) evaluates both the severity and extent of psoriasis lesions on four body regions: the scalp, arms, trunk, and legs. It assesses the percentage of body surface area affected by lesions (A=area score; 1=<10%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89%, 6=90-100%) and the severity of erythema (E), induration (I), and desquamation (D), each scored from 0 to 4.
  PASI scores range from 0 to 72, with higher scores indicating more severe disease.
ultrasonography | 1 day
  All participants included in the study will undergo sonographic examination using the Logiq 9 (GE, USA) ultrasound device and a high-frequency 7-12 MHz linear probe available in our clinic. The distance between the bilateral spina iliaca anterior superior and the upper pole of the patella of the participants' dominant and non-dominant extremities will be measured, and the distal 1/3 will be marked. The measurement will be taken in a seated upright position. Care will be taken to avoid compression during the measurement. After ensuring there is no compression in the subcutaneous fat tissue and muscle, an axial image will be recorded. The thickness of the subcutaneous fat tissue, vastus intermedius, rectus femoris, and total quadriceps will be measured three times, and the average of these measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Canan Dogan Tosun, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent; Tuba Güler, Assoc Prof, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy an Rehabilitation Hospital, Ankara, Bilkent-Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372